CLINICAL TRIAL: NCT04303039
Title: A Phase I Study to Investigate the Effects of Food on the Relative Bioavailability of a Tablet Formulation of ABP-671 in Healthy Subjects
Brief Title: Study to Investigate the Effects of Food on Relative Bioavailability of ABP-671 Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atom Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ABP-671-103
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Gout; Food-drug Interaction
MeSH Terms: conditions — Gout

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Single 1.0 mg dose of ABP-671 in the fasted state.
  Interventions: Drug: ABP-671
- Treatment B (Experimental): Single 1.0 mg dose of ABP-671 in the fed state, after a standardized breakfast.
  Interventions: Drug: ABP-671

INTERVENTIONS:
Drug: ABP-671 — ABP-671 Tablet 1.0 mg

SUMMARY:
This is a single center, open-label, single-dose, 2-way randomized crossover design in which 12 healthy subjects will be randomized to 1 of 2 treatment sequences (AB or BA). Treatments A and B will consist of single oral dose of tablet formulation (1.0 mg as 1 x 1.0 mg) in the fasted and fed state administered with approximately 240 mL of water. Each period will be separated by a washout interval of 4 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 60 years, inclusive
* Healthy
* Subjects must have the serum uric acid level at screening ≥ 3.7 mg/dL to ≤ 7.0 mg/dL for males, and ≥ 2.3 mg/dL to ≤ 6.0 mg/dL for females.
* Subjects must have a Body Mass Index (BMI) between 18 and 35 kg/m2 at screening (inclusive).
* Subjects must have a body weight of 50 kg or higher.
* Females must be non-pregnant and non-lactating
* Males must be surgically sterile, abstinent, or if engaged in sexual relations with a female partner of child-bearing potential, be using a condom with spermicide
* Subjects must have a CBC and platelet count within normal range
* Subjects must have normal blood chemistry
* Subjects must have a normal urinalysis
* Subjects meeting inclusion and exclusion criteria must have a renal ultrasound determined to be normal or non-clinically significant
* Subjects must have a normal estimated glomerular filtration rate
* Subjects must have a normal ECG
* Subjects must be able to comply with the study and follow-up procedures
* Subjects are able to understand the study procedures and risks involved and must provided signed informed consent to participate in the study

Exclusion Criteria:

* Subjects with any history or clinical manifestations of significant metabolic, hematological, pulmonary, including latent tuberculosis, cardiovascular, gastrointestinal including cholecystectomy, neurologic, hepatic, renal, urological, or psychiatric disorders.
* Subjects with prior history of bariatric surgery, intestinal resection, malabsorption, or celiac disease with an exception of subjects with appendectomy.
* Subjects who have any history or suspicion of kidney stones or evidence of renal stones or opacification with renal ultrasound prior to dosing on Day -1.
* Subjects who have any history of gout.
* Subjects who are positive for human immunodeficiency virus (HIV), Hepatitis B surface antigen, and/or Hepatitis C virus.
* Subjects who have used prescription drugs, over-the-counter drugs, or herbal remedies within 14 days screening period before Day 1 of study medication dosing. Females who have received hormone replacement therapy (HRT) within 14 days prior to dosing.
* Subjects who are positive for urine drug screening tests.
* Subjects who have undergone major surgery within 3 months prior to Day 1.
* Women who are pregnant or breastfeeding.
* Subjects who received any investigational test article within 5 half-lives or 30 days, whichever is longer, prior to Day 1 study medication dosing.
* Subjects who previously received ABP-671.
* Recent blood donation for more than 500 mL within 2 months of screening.
* Subjects who consumed Seville oranges- or grapefruit-containing foods or beverages within 7 days before Day 1 and during the entire study duration.
* Subjects with any condition that, in the judgment of the investigator, would place him/her at undue risk, or potentially compromise the results or interpretation of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
Plasma ABP-671 Concentration | 72 hours
  At times 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hrs.

SECONDARY OUTCOMES:
Serum Uric Acid Concentration | 72 hours
  At times 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hrs.
Serum Creatinine Concentration | 72 hours
  At times 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hrs.
Urine Uric Acid Concentration | 72 hours
  At times 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hrs.
Urine Creatinine Concentration | 72 hours
  At times 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hrs.

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron CPC, Inc., Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No